CLINICAL TRIAL: NCT00407225
Title: Phase 2a Study of 0.05% Difluprednate Ophthalmic Emulsion in the Treatment of Postoperative Inflammation After Cataract Surgery
Brief Title: Study of Difluprednate Ophthalmic Emulsion in the Treatment of Postoperative Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJE2079/2-01-PC
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2006-12-06 (Estimated); Status verified 2006-11

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

INTERVENTIONS:
Drug: Difluprednate Ophthalmic Emulsion

SUMMARY:
The purpose of this phase 2 study is to determine if difluprednate ophthalmic emulsion is effective in the treatment of postoperative inflammation.

DETAILED DESCRIPTION:
The objective is to assess the efficacy and safety of 0.002% and 0.05% difluprednate ophthalmic emulsions in patients with postoperative inflammation after cataract surgery (implantation of intraocular lens). In addition, the evaluation system for a future dose-finding phase III study of difluprednate ophthalmic emulsion will be established.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a mean postoperative (on the day of surgery or the day after surgery) flare intensity of 30 photon counts/msec
* Male and female patients aged 12 and <75 years who were able to accurately express their own symptoms
* Patients providing written informed consent prior to the start of the study
* Inpatients (patients were allowed to be discharged from the hospital during the study period)

Exclusion Criteria:

* Patients who did not meet any of the above inclusion criteria
* Patients receiving systemic administration, or topical application to the head or face (including instillation to the eyes) of any steroid, nonsteroidal anti-inflammatory drug, antiphlogistic enzyme, immunosuppressive drug or colchicine within 1 week prior to the start of the study treatment
* Patients with glaucoma or ocular hypertension (IOP: 21 mmHg)
* Patients with corneal abrasion or ulcer
* Patients with any viral keratoconjunctival disease, tuberculosus eye disease, fungal eye disease or bacterial eye disease
* Patients with diabetes who met any of the following criteria

  * HbA1C was 9.0% within 1 month prior to obtaining informed consent.
  * Proliferative diabetic retinopathy was present.
  * Rubeosis iridis was present.
* Patients with allergy to steroids
* Patients requiring the use of contact lens during the study period
* Women who were or might be pregnant
* Patients participating in another clinical study within 6 months prior to the start of the present study
* Patients sensitive to steroids (patients who previously experienced increased IOP after instillation of a steroid)
* Patients with a Grade 5 nuclear hardness as diagnosed according to Emery-Little classification
* Patients with fibrins or posterior rupture at baseline (F0)

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 1999-12; Study Completion 2000-10

PRIMARY OUTCOMES:
The flare intensity on Day 72 (F7) was compared with the baseline flare intensity (F0).
The ratios of the flare intensity on Day 1 (F1), that on Day 31 (F3) and that on Day 72 (F7) to
the baseline flare intensity (F0) (F1/F0, F3/F0 and F7/F0, respectively) were determined. Each
ratio was compared between the 0.002% and 0.05% difluprednate groups to identify when the
between-group difference in the effect of difluprednate became significant.

SECONDARY OUTCOMES:
The total score of anterior chamber signs (cells and protein) on Day 72 (S7) was compared
with the baseline total score (S0).
As the secondary efficacy evaluation, the ratios of the total score of anterior chamber signs
(cells and protein) on Day 1 (S1), that on Day 31 (S3) and that on Day 72 (S7) to the baseline
total score (S0) (S1/S0, S3/S0 and S7/S0, respectively) were determined. Each ratio was
compared between the 0.002% and 0.05% difluprednate groups to identify when the
between-group difference in the effect of difluprednate became significant.

CONTACTS AND LOCATIONS:
Overall Officials: Kanjiro Masuda, Study Chair — Director, Kanto Rosai Hospital; Director, Japanese Red Cross Medical Center